CLINICAL TRIAL: NCT04331054
Title: Protective Role of Inhaled Steroids for Covid-19 Infection
Acronym: INHASCO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 200394; 2020-001306-35 (EudraCT Number)
Record Dates: First submitted 2020-03-29; First posted 2020-04-02 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Covid-19 Infection; Hospitalization in Respiratory Disease Department
Keywords: Covid-19; Asthma; Inhaled steroids; Formoterol; Oxygen
MeSH Terms: conditions — COVID-19; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1: Usual practice (Active Comparator): arm will be follow during 30 days
  Interventions: Other: 1: Usual practice
- 2: Usual practice + SYMBICORT RAPIHALER (Experimental): Usual practice + SYMBICORT RAPIHALER 200/6 µg ( 2 puffs bid during 30 days)
  Interventions: Drug: 2: Usual practice + SYMBICORT RAPIHALER

INTERVENTIONS:
Drug: 2: Usual practice + SYMBICORT RAPIHALER — 2 puffs bid during 30 days by inhalation
  Arms: 2: Usual practice + SYMBICORT RAPIHALER
Other: 1: Usual practice — Usual practice
  Arms: 1: Usual practice

SUMMARY:
We hypothesize that inhaled steroid therapy and long acting beta 2 adrenergic agonist, widely prescribed in asthma patients, may also have a local protective effect against coronavirus infection, even in patients without asthma.

The primary purpose is To compare time to clinical improvement in patients receiving standard of care associated to the combination budesonide/formoterol or standard of care only.

Time (in days) to clinical improvement is defined as the time from randomization to an improvement of two points (from the status at randomization) on a seven-category ordinal scale or live discharge from the hospital, whichever came first within 30 days.

DETAILED DESCRIPTION:
D1 inclusion / randomization visit:

Patients who meet the eligibility criteria and whose infection with Covid-19 has been confirmed within 48 hours will be included in the respiratory diseases department by the pneumologist investigator.

Patients will be randomized either to the control group or to the intervention group. For interventional patients, trial treatment (SYMBICORT RAPIHALER 200/6 µ) will begin within 12 hours.

Follow-up period (D2 to D29) and end of study visit (D30):

Throughout their hospital stay, patients will be followed in accordance with the practice of the service.

During hospitalization, investigators are free to decide for antibiotics, steroids, anti viral drugs, hydroxychloroquine and oxygen support management in accordance with local practice. None of the laboratory tests are made for the study. They are usually performed in patients hospitalized for acute respiratory infection.

Interventional patient will also be treated with SYMBICORT RAPIHALER 200/6 µg (2 puffs 2 times a day).

In the event that the patient is discharged from hospital before the end of his participation, he will be contacted by phone on D30 in order to obtain information concerning the period outside hospitalization

ELIGIBILITY:
Inclusion criera :

* Patient ≥ 18 years old and ≤ 75 years old
* Laboratory proved infection by COVID-19 by RT-PCR on a respiratory biological sample within 2 days
* Hospitalization is required according to current local recommendations
* Patient affiliated to a social security regime
* Patient able to give free, informed and written consent

Exclusion criteria :

* Oxygen flow rate >8l/min at inclusion
* Current treatment with any inhaled steroid (any other form of steroid administration does not exclude the patient)
* Intensive care unit is required for the patient (based on investigator judgement)
* Patient with cognitive impairment which do not guarantee proper use of the treatment by the patient himself
* Pregnant (positive β-HCG at inclusion) or breastfeeding women
* Participation in another interventional drug study involving human participants and concerning COVID-19 infection or being in the exclusion period of a previous study involving human participants
* Contraindications to the treatments (history of hypersensitivity)
* Patient admitted for isolation, for social reason or due to comorbidities without gravity sign
* Long-term patient treated with digitalis, disopyramide, procainamide or phenothiazine that could lengthen the QT space

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Time (in days) to clinical improvement within 30 days after randomization | within 30 days
  Time (in days) to clinical improvement is defined as the time from randomization to an improvement of two points (from the status at randomization) on a seven-category ordinal scale or live discharge from the hospital, whichever came first within 30 days.
  The seven-category ordinal scale consisted of the following categories:
  1. Not hospitalized with resumption of normal activities
  2. Not hospitalized, but unable to resume normal activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, requiring nasal high-flow oxygen therapy, non-invasive mechanical ventilation, or both;
  6. Hospitalized, requiring ECMO, invasive mechanical ventilation, or both
  7. Death.
  These parameters will be evaluated daily during hospitalization.

SECONDARY OUTCOMES:
Mortality rate at D30 | At day30
Time (in days) from randomization to death | up to 30 days after randomization
Number of days alive outside ICU within 30 days | At day30
Number of days alive free of invasive or non-invasive ventilation within 30 days | At day30
Number of days alive with oxygen therapy within 30 days | At day30
Maximal oxygen rate within 30 days | At day30
Difference between PaO2/FiO2 ratio at randomization and at Day 7 (or at the time of stopping oxygen therapy or discharge if occurs before Day 7) | at Day 7
Number of days alive outside hospital within 30 days | at Day 30
Use of antibiotics for respiratory (proved or suspected) infection within 30 days | at Day 30
Difference between CRP levels at randomization and at Day 7 (or at the time of discharge if occurs before Day 7) | at Day 7
Safety outcomes included events that occurred during treatment, serious adverse events, and premature discontinuation of treatment. | up to 30 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Camille TAILLE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat - Service de Pneumologie, Paris, France